CLINICAL TRIAL: NCT01740245
Title: Antisepsis Regimen in the Surgical Treatment of Human Papilloma Virus Generated Cervical Lesions: Polyhexamethylene Biguanide Versus Chlorhexidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: CHX-PHMB
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-06

CONDITIONS: Antisepsis Regimen After Surgical Treatment of HPV Infected Lesions
Keywords: Laser therapy; Cervical lesions; Polyhexamethylene biguanide; Chlorhexidine

ARMS (2):
- Chlorhexidine (Active Comparator)
  Interventions: Device: Chlorhexidine vaginal suppositories
- Polyhexamethylene biguanide (Experimental)
  Interventions: Device: Polyhexamethylene biguanide vaginal suppositories

INTERVENTIONS:
Device: Chlorhexidine vaginal suppositories
  Arms: Chlorhexidine
Device: Polyhexamethylene biguanide vaginal suppositories
  Arms: Polyhexamethylene biguanide

SUMMARY:
Treatments for the macroscopic or pathologic lesions caused by HPV infection can be classified as topical, surgical, destructive, or immunomodulatory. Post surgical treatments generally consist of analgesic, anti-inflammatory and topical antimicrobial agents to reduce the risk of local infections.

The aim of this study is to compare the efficacy and safety of polyhexamethylene biguanide-based vaginal suppositories to a similar chlorhexidine-based treatment, in the post recovery regimen after surgical treatment of cervical lesions.

Women who underwent to CO2 laser therapy for cervical lesions are randomly assigned to receive 10 days of antiseptic treatment with chlorhexidine digluconate vaginal suppositories, or polyhexamethylene biguanide vaginal suppositories (Monogin® / BiguanelleTM vaginal suppositories, Lo.Li.Pharma, Italy). A weekly follow-up check was performed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* positive colposcopy examination
* positive Papanicolaou smear
* pathological biopsy
* physical ablation by CO2 laser therapy for a number of lesions included between 3 and 5

Exclusion Criteria:

* pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Bacterial vaginosis | After three weeks by the day of the laser treatment
  Diagnosis of eventual bacterial infection is performed according to Amsel's criteria
Change from baseline bleeding at 6 weeks | At weekly intervals by the day of laser treatment
  Visual scoring was assessed depending on the grade of the defect (from 1 to 3)
Change from baseline healing process at 6 weeks | At weekly intervals by the day of laser treatment
  Visual scoring for healing is assessed depending on the grade of the defect (from 1 to 3)
Change from baseline irritation status at 6 weeks | At weekly intervals by the day of laser treatment
  Visual scoring for irritation is assessed depending on the grade of the defect (from 1 to 3)
Bacterial vaginosis | After six weeks by the day of laser treatment
  Diagnosis is performed according to the Amsel's criteria

CONTACTS AND LOCATIONS:
Locations (1):
- AGUNCO, Rome, Italy

REFERENCES:
- [Background] Wiley DJ, Douglas J, Beutner K, Cox T, Fife K, Moscicki AB, Fukumoto L. External genital warts: diagnosis, treatment, and prevention. Clin Infect Dis. 2002 Oct 15;35(Suppl 2):S210-24. doi: 10.1086/342109. PMID 12353208
- [Background] Kaehn K. Polihexanide: a safe and highly effective biocide. Skin Pharmacol Physiol. 2010;23 Suppl:7-16. doi: 10.1159/000318237. Epub 2010 Sep 8. PMID 20829657
- [Background] Koburger T, Hubner NO, Braun M, Siebert J, Kramer A. Standardized comparison of antiseptic efficacy of triclosan, PVP-iodine, octenidine dihydrochloride, polyhexanide and chlorhexidine digluconate. J Antimicrob Chemother. 2010 Aug;65(8):1712-9. doi: 10.1093/jac/dkq212. Epub 2010 Jun 15. PMID 20551215
- [Background] Muller G, Kramer A. Biocompatibility index of antiseptic agents by parallel assessment of antimicrobial activity and cellular cytotoxicity. J Antimicrob Chemother. 2008 Jun;61(6):1281-7. doi: 10.1093/jac/dkn125. Epub 2008 Mar 25. PMID 18364400